CLINICAL TRIAL: NCT06581354
Title: The Impact of Provisionalization Using Glass Fiber Reinforced Composite on Patient Satisfaction and Prosthetic Complications in Maxillary Implant-Supported Arches Restored by Definitive Pekkton Frameworks
Brief Title: GFRC Enhance Patient Satisfaction and Reduce Complications in Maxillary Implants With Pekkton Frameworks
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana Mohamed Abdelhamed Shehata, principal investigator (assistant lecturer of prosthodontics), Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2 1 24
Record Dates: First submitted 2024-08-19; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Edentulous Alveolar Ridge

STUDY DESIGN:
Intervention Model Description: Group I: Intervention will be treated using a glass fiber composite as a temporary framework followed by PEKKTON definitive framework.
  Group II: Controls will be treated using PEKKTON definitive framework (no provisionalization).
Who Masked: Outcomes Assessor
Masking Description: The study will be based on different technical procedures for the fabrication of the frameworks. Since these differences are visible, the operator and the technician involved in the study as well as the outcome assessor cannot be blinded. But the statistician and patients will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- no provisional prosthesis, pekkton is a definitive framework. (Active Comparator): Implant-supported, full-arch maxillary prosthesis utilizing 6 implants, for constructing PEKKTON framework without provisionalization
  Interventions: Procedure: PROVISIONALIZATION
- Glass fiber composite framework for provisionalization then pekkton framework. (Experimental): Implant-supported full arch maxillary provisional prosthesis protocol utilizing 6 implants for constructing a resin glass fiber composite framework followed by a definitive PEKKTON framework.
  Interventions: Procedure: PROVISIONALIZATION

INTERVENTIONS:
Procedure: PROVISIONALIZATION — glass fiber composite as a temporary framework followed by PEKKTON definitive framework.

SUMMARY:
This study aims to evaluate the effect of provisionalization with a glass fiber composite framework on patient satisfaction and prosthetic complications before the insertion of a definitive PEKKTON framework when used under the screw-retained maxillary implant-supported prostheses at a one-year follow-up period.

DETAILED DESCRIPTION:
1. Patient grouping:

   Group I: (intervention) Patients obtained an Implant-supported full arch maxillary provisional prosthesis protocol utilizing 6 implants for constructing a resin glass fiber composite framework followed by a definitive PEKKTON framework.

   Group II: (control) patients obtained an Implant-supported, full arch maxillary definitive prosthesis utilizing 6 implants, for constructing PEKKTON framework without provisionalization.
2. Preparation of a scan appliance:

   * The patient's denture will be used as a scan appliance by the addition of radiopaque material to act as radiopaque markers over the polished surfaces of the prosthesis in a staggered pattern at different levels to the occlusal plane on the buccal, labial, and palatal flanges of the denture.
   * Double scan protocol will be used in our study in which a cone beam conventional tomography (CBCT) images will be produced for each case. The first scan will be taken for the maxilla while the patient is wearing the maxillary denture with the radiopaque markers and biting over cotton rolls, the other scan is for the modified maxillary denture.
   * Computer software (BlueSky Bio) was used to overlap the two scans on each other where the final file contained reformatted images in 3D bone model, and 3D radiographic modified denture guide model to construct the surgical guide.
3. Virtual planning, surgical guide fabrication, and Implant placement

   * The implant planning will be done using the BlueSky Bio software. The scan of the maxillary denture will be superimposed over that of the maxillary arch scan, using points over the radiopaque marker as alignment points, for proper orientation of the scan appliance.
   * 6 Implant planning {(3.7x12) for the anterior segment and (4x10) for the posterior segment} will be placed in areas with high bone quality and quantity of bone and will be distributed according to AP spread.
   * A surgical guide will be planned and then the 3D virtual guide will be exported as STL file to the 3D printing machine. The surgical guide will be fixed in place using three fixation screws; with an adequate distance from the planned implant drilling sites, two screws placed in the buccal shelf area on both sides, and one screw in the midline to achieve a tripoding position.
   * The 3D surgical guide will be provided with metal sleeves corresponding to the virtually planned drilling sites with the precise depth, angulation, mesiodistal and buccolingual positioning of each implant as planned during the computer simulation for accurate placement of the implants' osteotomies. The osteotomies will be drilled, and implants will be inserted.
   * The multi-unit abutments will be placed over the dental implants. The denture will be relieved around the abutments and picked up by soft liner.
   * All patients will be instructed about oral hygiene measures, a soft diet for 4 weeks after surgery, and antimicrobial prophylaxes (amoxicillin 500mg twice daily for 5 days starting 1 hour before surgery). Postsurgical analgesic treatment will be performed with ibuprofen 600mg twice daily.
4. Prosthetic procedures: After 1 Month:

   * Group one: will be rehabilitated by using a glass fiber composite as a temporary framework followed by PEKKTON definitive framework.

Framework fabrication:

* The glass fiber composite framework and PMMA teeth will be digitally designed according to implant location, crown height space, occlusion, and opposing complete denture with the help of scan appliance wax up.
* The framework will be placed over the multi-unit abutments intraorally, picked up on the cylinder and. The occlusion of printed teeth by PMMA will be checked and then cemented with the framework. Then the whole assembly will be removed from the patient's mouth.
* After one month, the printed composite framework with the printed PMMA teeth will be screwed intraorally.
* After four months of temporization, the definitive PEKKTON will be re-milled from the same scan and delivered to the patients with the milled teeth.
* These frameworks will be milled, the passive fit will be checked between frameworks and multi-unit abutments, and the occlusion of printed teeth by PMMA will be checked and tried intra-orally. If the try-in is accepted, the assigned material (PMMA) will be milled and assembled to the framework.
* Group two: patients obtained an Implant-supported, full-arch maxillary prosthesis utilizing 6 implants, for constructing PEKKTON framework without provisionalization.

A. Digital impressions Scan bodies will be tightened onto the multi-unit abutments and an intraoral digital impression will be made using an IOS system after one month of implant insertion.

B. Verification jigs fabrication (digitally) The milled PMMA jig will be constructed and checked for passive seating on implants by verifying proper contact at the PMMA jig interface and the multi-unit abutments.

C. Framework fabrication:

* The (PEKKTON) frameworks and teeth will be digitally designed according to implant location, crown height space, occlusion, and opposing dentition with the help of scan appliance wax up.
* The frameworks will be milled with the final material (PEKKTON) and teeth will be printed with temporary material (PMMA).
* First, the passive fit will be checked between frameworks and multi-unit abutments, and the occlusion of printed teeth by PMMA will be checked and tried intra-orally.
* Accordingly, if the try-in is accepted, the assigned material (PMMA) will be milled and assembled to the framework.
* Glass fiber composite (Trilor fiber disc) with 98mm diameter and 16mm height, bio-Loren company, made in Italy, 21047 saronno (va)Italy.
* PEKKTON ivory, High-performance polymer, Cendres +métaux

ELIGIBILITY:
Inclusion Criteria:

* a. Completely edentulous patients with Angle's Class I maxillomandibular relationship b. Age ranges from 40 to 65 years old. c. Adequate zone of keratinized attached mucosa (≥ 8mm) over the maxillary crest.

  d. Absence of any medical disorder that could complicate the surgical phase or affect osseointegration.

  e. The patient must have enough bone height for implants, a minimum length of bone f. 12 mm, and a minimum diameter of bone 6 mm. g. Patients with good oral hygiene. h. Complete denture wearer. i. Adequate interarch space for screw-retained prosthesis. j. Absence of any intra-oral pathological condition.

Exclusion Criteria:

- a. Patients with recent extraction (less than three months). b. Patients with an inflamed ridge or candida infection c. Patients with the flabby ridge. d. Para functional habits. e. Cancer patients receiving chemotherapy and/or radiotherapy. f. Patients with uncontrolled diabetes, assessed by measuring glycosylated hemoglobin (HbA1c ≥ 7) g. Potentially uncooperative patients who are not willing to go through the proposed interventions.

h. Moderate-to-heavy daily smokers (more than ten per day)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | one year
  During the 12-month follow-up period as follows (3 months after delivery, 6 months after delivery, and 12 months after delivery), Patient satisfaction for Implant-supported screw-retained full arch maxillary provisional prosthesis with early loading protocol utilizing 6 implants for constructing a resin glass fiber composite followed by (PEKKTON) framework will be registered and calculated by Questionnaire

SECONDARY OUTCOMES:
prosthetic complications | one year
  During the 12-month follow-up period as follow( 3 months after delivery, 6 months after delivery, and 12 months after delivery), Prosthetic complications for Implant-supported screw-retained full arch maxillary provisional prosthesis with early loading protocol utilizing 6 implants for constructing a (PEKKTON) framework will be registered and calculated according to the following events: screw loosening of the abutment, screw loosening of the prosthesis, fracture of the screw of the abutment, fracture of the screw of the prosthesis, abutment fracture, framework fracture, fracture of acrylic resin denture, loss of cover of access hole, prosthetic teeth fracture and remake of the prosthesis, occlusal discrepancies, maxillary and mandibular denture relining if needed, pain.

CONTACTS AND LOCATIONS:
Overall Officials: rana shehata, phd, Principal Investigator — faculty of dentistry Cairo university -Egypt

IPD SHARING:
Plan to Share IPD: No
sharing the main point of methodology and the final results